CLINICAL TRIAL: NCT03117244
Title: A Protocol for Muscular Foot Strengthening On a Capacity to Control the Deformation of the DOT Plantar Medial
Brief Title: The Effectiveness of a Protocol for Muscular Foot Strengthening On a Capacity to Control the Deformation of the DOT Plantar Medial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Claudio Cazarini Junior, Physical therapist, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 62766716.4.0000.5479
Record Dates: First submitted 2017-04-10; First posted 2017-04-17 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Foot Diseases
MeSH Terms: conditions — Foot Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise Group (Experimental)
  Interventions: Other: Exercise for Foot Strengthening
- Exercise and NMES Group (Active Comparator)
  Interventions: Other: Exercise for Foot Strengthening and Electrostimulation
- Control Group (No Intervention)

INTERVENTIONS:
Other: Exercise for Foot Strengthening — Stabilization exercises of the longitudinal arch of the foot
  Arms: Exercise Group
Other: Exercise for Foot Strengthening and Electrostimulation — Exercise for the Strengthening of the Foot associated with Electrostimulation
  Arms: Exercise and NMES Group

SUMMARY:
The human foot allows to perform several functions, rather than providing a Static support for the body, the foot acts dynamically in walking and Movement of the body, requiring adequate biomechanics responsible for Maintenance and posture of the body and harmonic distribution of plantar pressure.

One of the most important structures for this control is the medial plantar vault (MPA), an important structure in the absorption of impact and essential for the function Foot. The deformation of the MPA in the gait support phase absorbs the Energy and propels the limb, to perform this biomechanical function the MPA must Stable from the anatomical point of view, which is conferred by the bone architecture and But also by the performance of the intrinsic and extrinsic musculature of the Feet. The fall of the MPA, decreases the stability of the foot, limits its biomechanical function,

Besides being a risk factor for the development of pathologies such as:

Tendinopathy of the calcaneus tendon and plantar fasciitis. Various Intrinsic Muscles And extrinsic have the function of stabilizing the foot and the MPA, being the main Extrinsic muscles: the posterior tibial, the flexor long of the hallux and the fingers. The Muscles when activated increase the height and decrease the Length of the MPA. Several methods are used to evaluate ALM, such as (AN), Feiss line (LF) and MPA angle (MPAH), in addition to the Baropodometry, which is used to evaluate dysfunctions in the feet, with the principle of Map the pressure of the plantar surface in a static and dynamic way. Based In this information, this study aims to evaluate the influence of the Strengthening of the intrinsic and extrinsic muscles of the feet, for the Of MPA in asymptomatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18 and 40,
* Seeders (do not practice physical activity regularly)
* No previous injuries to the feet and ankles,
* 12 months without lesions in lower members,
* Without deformities in APM,
* Such as, rigid planar foot
* No history of neurological changes

Exclusion Criteria:

* Individuals who practice physical activities regularly,
* History of pain in the feet,
* Have suffered fractures in the lower limbs,
* Muscular and articular lesions of Lower members in 12 months, -
* Flat foot,
* Valgus of calcaneus above 10º
* History of neurological changes or surgical procedure performed on lower limbs

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Measurements of the medial longitudinal arch | 6 weeks
  Navicular height Angle of the medial longitudinal arch Feiss line

CONTACTS AND LOCATIONS:
Locations (1):
- Claudio Cazarini Júnior, São Paulo, São Paulo, Brazil